CLINICAL TRIAL: NCT01000831
Title: PCIRN Evaluation of Pandemic H1N12009 Influenza Vaccine After One andTtwo Doses in Young Children
Brief Title: Rapid Evaluation of Pandemic H1N1 Influenza Vaccines in Young Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); PHAC/CIHR Influenza Research Network (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H09-02749
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Influenza
Keywords: vaccine; influenza; H1N1 influenza vaccine; influenza vaccine; Arepanrix
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adjuvanted Arepanrix 2 doses (Active Comparator): Two doses of adjuvanted H1N1 Arepanrix vaccine given 3 weeks apart
  Interventions: Biological: adjuvanted Arepanrix

INTERVENTIONS:
Biological: adjuvanted Arepanrix — Two doses of adjuvanted Arepanrix vaccine given 3 weeks apart
  Other Names: Influenza vaccine

SUMMARY:
The purpose of this study is to compare the safety and effectiveness (immune response) to one or two doses of adjuvanted H1N12009 influenza vaccine in young children. An adjuvant is an additive that can boost the immune response. The study will enroll 300 children (ages 6-35 months). Participants will receive 2 doses of adjuvanted H1N12009 vaccine 3 weeks apart. Study procedures include: medical history, blood samples and completing a memory aid. Participants will be involved in study related procedures for approximately 6 weeks.

DETAILED DESCRIPTION:
The goal of this study is to determine if one or two doses of the H1N12009 influenza vaccine are needed in young children, a population group at high risk of influenza infection and subsequent hospitalization.

The objectives of this study are two-fold:

1. To compare the safety and immunogenicity of 1 and 2 doses of adjuvanted H1N12009 influenza vaccine in children 6-35 months of age.
2. To conduct the trial soon after the vaccines become available and share the observations with health officials and the public as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided for the subject by a parent or legal guardian
* Children age 6-35 months

Exclusion Criteria:

* Allergies to eggs, thimerosal, gentamicin sulphate or latex
* Life-threatening reaction to previous Flu vaccine
* Bleeding disorder
* Pregnancy
* Receipt of blood or blood products in past 3 months
* Chronic illness that could interfere with trial participation
* Compromised immune system
* Previous lab-confirmed H1N12009 infection
* Receipt of H1N12009 vaccine
* Receipt of Seasonal Influenza vaccine since March 2009

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 167 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety and immunogenicity of one and two doses Arepanrix | Day 7 and Day 21 post vaccination measured at day 42
  To compare the safety and immunogenicity of one and two doses of adjuvanted H1N12009 pandemic vaccine in children 6-35 months of age
Rapid Trial | Day 42
  To conduct this trial soon after the vaccines become available and share observations with health officials and the public as soon as possible

CONTACTS AND LOCATIONS:
Overall Officials: David Scheifele, MD, Principal Investigator — University of British Columbia; Marc Dionne, MD, Study Director — Unité de Recherche en Santé Publique (CHUQ); Brian Ward, MD, Principal Investigator — McGill University Health Center - Vaccine Study Center; Joanne Langley, MD, Study Director — Canadian Center for Vaccinology, Dalhousie University; Otto Vanderkooi, MD, Study Director — Alberta Children's Hospital, University of Calgary; Simon Dobson, MD, Study Director — University of British Columbia
Locations (6):
- Canada (6):
  - Alberta Children's Hospital, University of Calgary, Calgary, Alberta
  - Child and Family Research Institute, Vancouver, British Columbia
  - Vaccine Evaluation Center, University of British Columbia, Vancouver, British Columbia
  - Canadian Center for Vaccinology, Dalhousie University, Halifax, Nova Scotia
  - McGill University Health Center - Vaccine Study Center, Montreal, Quebec
  - Unité de Recherche en Santé Publique (CHUQ), Québec, Quebec

REFERENCES:
- [Result] Scheifele DW, Ward BJ, Dionne M, Vanderkooi O, Langley JM, Dobson S, Li Y, Law B, Halperin SA; Public Health Agency of Canada/Canadian Institutes of Health Research Influenza Research Network (PCIRN) Rapid Trials Investigators. Evaluation of adjuvanted pandemic H1N1(2009) influenza vaccine after one and two doses in young children. Pediatr Infect Dis J. 2011 May;30(5):402-7. doi: 10.1097/INF.0b013e3182068f33. PMID 21178654